CLINICAL TRIAL: NCT02003144
Title: A Phase III, Open-label, Extension Trial of ECU-NMO-301 to Evaluate the Safety and Efficacy of Eculizumab in Patients With Relapsing Neuromyelitis Optica (NMO)
Brief Title: An Open Label Extension Trial of Eculizumab in Relapsing NMO Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECU-NMO-302; 2013-001151-12 (EudraCT Number)
Record Dates: First submitted 2013-11-18; First posted 2013-12-06 (Estimated); Results first posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-07

CONDITIONS: Neuromyelitis Optica; Neuromyelitis Optica Spectrum Disorder
Keywords: Long-term safety study; Extension trial; Eculizumab; Neuromyelitis Optica Spectrum Disorder; Devic's disease; Transverse Myelitis; Optic Neuritis; Relapse; NMO-IgG; CNS Autoimmune Disorders; Demyelinating Disorders
MeSH Terms: conditions — Neuromyelitis Optica; Myelitis, Transverse; Optic Neuritis; Recurrence; Demyelinating Diseases | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eculizumab (Experimental): Eculizumab intravenous infusion every two weeks.
  Interventions: Biological: eculizumab

INTERVENTIONS:
Biological: eculizumab
  Other Names: Soliris

SUMMARY:
The purpose of this study is to determine whether eculizumab long-term use is safe and effective in patients with relapsing NMO.

DETAILED DESCRIPTION:
This study is an open label extension study to confirm the long term safety and efficacy of eculizumab in subjects with relapsing NMO who have completed the initial double-blind, randomized, placebo-controlled trial ECU-NMO-301.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patient completed the ECU-NMO-301 trial
2. Patient has given written informed consent

Key Exclusion Criteria:

1. Patients who have withdrawn from the ECU-NMO-301 trial as a result of an AE related to trial drug
2. Female patients who are pregnant, breastfeeding, or intend to conceive during the course of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (69):
- United States (19):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - The Research Center of Southern California, Oceanside, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami McKnight Brain Institute, Miami, Florida
  - Neurological Services of Orlando, Orlando, Florida
  - Allied Physicians Inc. of Fort Wayne, Fort Wayne, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Baptist Health Lexington, Nicholasville, Kentucky
  - Johns Hopkins University Medical Center, Baltimore, Maryland
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Multiple Sclerosis Comprehensive Care Center NYU Langone Medical Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Ohio Health Reserach Institute, Columbus, Ohio
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Multiple Sclerosis Treatment Center of Dallas, Dallas, Texas
  - The University of Texas Health Science, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
- Argentina (4):
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Fundacion Rosarina de Neuro Rehabilitacion, Rosario, Santa Fe Province
  - Hospital General de Agudos Juan Antonio Fernandez, Ciudad Autonoma, Buenos Aires
  - Hospital General de Agudos Dr. J. M. Ramos Mejia, Ciudad Autonoma, Buenos Aires,
- Australia (2):
  - Brain and Mind Research Institute, Camperdown, New South Wales
  - St. Vincent's Hospital, Fitzroy, Victoria
- The Ottawa Hospital, Ottawa, Ontario, Canada
- Fundacion Cardiovascular de Colombia, Floridablanca, Santander Department, Colombia
- Clinical Hospital Centre Zagreb, Zagreb, Croatia
- Czechia (2):
  - VFN v Praze, Prague
  - Krajska zdravotni, a.s. - Nemocnice, Teplice
- Århus Universitetshospital, Aarhus, Denmark
- Germany (4):
  - University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg
  - Neurologische Klinik und Poliklinik, Munich, Bavaria
  - University Hospital Heinrich Heine University, Düsseldorf, North Rhine-Westphalia
  - Universitaetsmedizin Rostock, Rostock
- Prince of Wales Hospital, Shatin, Hong Kong
- Italy (4):
  - Policlinico di Catania, Catania
  - Azienda Ospedaliera Universitaria, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Rome
- Japan (7):
  - Chiba University Hospital, Chiba, Chiba
  - Hyogo College of Medicine Hospital, Nishinomiya-shi, HyogoKen
  - Kyoto Min-iren Chuo Hospital, Kyoto, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Yamaguchi University Hospital, Ube-shi, Yamaguchi
  - Kyushu University Hospital, Fukuoka
  - National Center Hospital, NCNP, Tokyo
- Malaysia (2):
  - Hospital Umum Sarawak, Kuching, Sarawak
  - Hospital Kuala Lumpur, Kuala Lumpur
- Russia (4):
  - Republican Clinical Hospital for Rehabilitation of Healthcare Ministry of Republic of Tatarstan, Kazan'
  - SBEI "Krasnoyarsk SMU n.a. Prof. V.F. Voyno-Yasenetsky", Krasnoyarsk
  - Federal State Budget Institution of Healthcare - Siberian District Medical Center of FMBA of Russia, Novosibirsk
  - SEIHPE "Rostov SMU of MoH of RF", Rostov-on-Don
- South Korea (5):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul University National Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
- Spain (3):
  - Hospital de Cruces, Barakaldo, Bizkaia
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Clinico San Carlos, Madrid
- Cheng Hsin General Hospital, Taipei, Taiwan
- Thammasat University Hospital, Pathum Thani, Thailand
- Turkey (Türkiye) (5):
  - Hacettepe University Medical Faculty, Ankara
  - Trakya University Medical Faculty, Edirne
  - Dokuz Eylul University Medicine Faculty, Izmir
  - Kocaeli University Medical Faculty, Kocaeli
  - Ondokuz Mayis Univ. Med. Fac., Samsun
- The Walton Centre, Liverpool, United Kingdom

REFERENCES:
- [Background] Pittock SJ, Lennon VA, McKeon A, Mandrekar J, Weinshenker BG, Lucchinetti CF, O'Toole O, Wingerchuk DM. Eculizumab in AQP4-IgG-positive relapsing neuromyelitis optica spectrum disorders: an open-label pilot study. Lancet Neurol. 2013 Jun;12(6):554-62. doi: 10.1016/S1474-4422(13)70076-0. Epub 2013 Apr 26. PMID 23623397
- [Derived] Pittock SJ, Fujihara K, Palace J, Berthele A, Kim HJ, Oreja-Guevara C, Nakashima I, Levy M, Shang S, Yountz M, Miller L, Armstrong R, Wingerchuk DM; PREVENT Study Group. Eculizumab monotherapy for NMOSD: Data from PREVENT and its open-label extension. Mult Scler. 2022 Mar;28(3):480-486. doi: 10.1177/13524585211038291. Epub 2021 Sep 9. PMID 34498507
- [Derived] Kim HJ, Nakashima I, Viswanathan S, Wang KC, Shang S, Miller L, Yountz M, Wingerchuk DM, Pittock SJ, Levy M, Berthele A, Totolyan N, Palace J, Barnett MH, Fujihara K; PREVENT Study Group. Eculizumab in Asian patients with anti-aquaporin-IgG-positive neuromyelitis optica spectrum disorder: A subgroup analysis from the randomized phase 3 PREVENT trial and its open-label extension. Mult Scler Relat Disord. 2021 May;50:102849. doi: 10.1016/j.msard.2021.102849. Epub 2021 Feb 20. PMID 33676197

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed Study ECU-NMO-301 (NCT01892345) were eligible to participate in Study ECU-NMO-302. This is an open-label study in which all participants were administered intravenous eculizumab. However, to maintain the blind of Study ECU-NMO-301, all participants underwent a 4-week Blind Induction Phase before entering the Open-label Maintenance Phase.
Groups:
- Placebo/Eculizumab: Blind Induction Phase: Participants who had received blinded treatment with placebo in Study ECU-NMO-301 were administered eculizumab (900 milligrams [mg]) plus matching placebo via intravenous (IV) infusion on Day 1 and Weeks 1 through 3. Open-Label Maintenance Phase: Participants received open-label eculizumab (1200 mg) via IV infusion every 2 weeks starting at Week 4 and continued for up to 6.5 years.
- Eculizumab/Eculizumab: Blind Induction Phase: Participants who had received blinded treatment with eculizumab in Study ECU-NMO-301 were administered eculizumab (1200 mg) via IV infusion on Day 1 and Week 2 and placebo at Weeks 1 and 3. Open-Label Maintenance Phase: Participants received open-label eculizumab (1200 mg) via IV infusion every 2 weeks starting at Week 4 and continued for up to 6.5 years.
Period: Blind Induction Phase
Arm/Group | Placebo/Eculizumab | Eculizumab/Eculizumab
Started | 41 | 78
Received at Least 1 Dose of Study Drug | 41 | 78
Completed | 41 | 78
Not Completed | 0 | 0
Period: Open Label Maintenance Phase
Arm/Group | Placebo/Eculizumab | Eculizumab/Eculizumab
Started | 41 | 78
Received at Least 1 Dose of Study Drug | 41 | 78
Completed | 32 | 64
Not Completed | 9 | 14
Not completed — Other than specified | 2 | 4
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Pregnancy | 0 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Extension Full Analysis Set consisted of all participants who had received at least 1 dose of eculizumab in Study ECU-NMO-302 and have a post-IP-infusion efficacy assessment.
Groups:
- Placebo/Eculizumab: Blind Induction Phase: Participants who had received blinded treatment with placebo in Study ECU-NMO-301 were administered eculizumab (900 mg) plus matching placebo via IV infusion on Day 1 and Weeks 1 through 3. Open-Label Maintenance Phase: Participants received open-label eculizumab (1200 mg) via IV infusion every 2 weeks starting at Week 4 and continued for up to 6.5 years.
- Total: Total of all reporting groups
Arm/Group | Placebo/Eculizumab | Eculizumab/Eculizumab | Total
Number analyzed (Participants) | 41 | 78 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (13.82) | 46.6 (13.77) | 46.4 (13.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 74 | 110
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 11 | 13
  Not Hispanic or Latino | 37 | 63 | 100
  Unknown or Not Reported | 2 | 4 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 13 | 32 | 45
  Black or African American | 7 | 3 | 10
  White | 21 | 40 | 61
  Other | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Treatment-emergent adverse events (TEAEs) were defined as an AE with onset on or after the first study drug dose in Study ECU-NMO-302. A serious adverse event (SAE) was defined as an untoward medical occurrence that at any dose either results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline up to end of study (up to 6.5 years)
Population: The Extension Safety Set consisted of all participants who had received at least 1 dose of eculizumab in Study ECU-NMO-302.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Eculizumab | Eculizumab/Eculizumab
Number analyzed (Participants) | 41 | 78
Participants
  TEAEs | 41 | 70
  SAEs | 14 | 26

2. Primary Outcome: Number of Participants With At Least 1 Post Baseline Columbia-Suicide Severity Rating Scale (C-SSRS) Assessment (Suicide-Related Thoughts or Behaviours) Abnormality
Description: The C-SSRS is a validated questionnaire to capture occurrence, severity, and frequency of suicide-related thoughts and behaviours, and has a binary response (yes/no). Suicidal Ideation: a "yes" answer to any one of 5 suicidal ideation questions: Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Planned) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; and Active Suicidal Ideation with Specific Plan and Intent. Suicidal Behaviour: a "yes" answer to any of 5 suicidal behaviour questions: Preparatory Acts or Behaviour, Aborted Attempt, Interrupted Attempt, Actual Attempt (non-fatal), and Completed Suicide. Suicidal Ideation or Behaviour: a "yes" answer to the following question: Self-injurious behaviour without suicidal intent.
Time Frame: Baseline up to end of study (up to 6.5 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Eculizumab | Eculizumab/Eculizumab
Number analyzed (Participants) | 41 | 78
Participants
  Suicidal Ideation | 4 | 5
  Suicidal Behavior | 0 | 1
  Suicidal Ideation or Behavior | 4 | 5

3. Primary Outcome: Number of Participants With An On-trial Relapse as Determined by The Treating Physician
Description: An On-trial Relapse was defined as a new onset of neurologic symptoms or worsening of existing neurologic symptoms with an objective change (clinical sign) on neurologic examination that persisted for more than 24 hours as confirmed by the treating physician.
Time Frame: Baseline up to end of study (up to 6.5 years)
Population: The Extension Full Analysis Set consisted of all participants who had received at least 1 dose of eculizumab in Study ECU-NMO-302 and had a post-IP-infusion efficacy assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Eculizumab | Eculizumab/Eculizumab
Number analyzed (Participants) | 41 | 78
Participants | 5 | 8

4. Primary Outcome: On-Trial Annualized Relapse Rate (ARR) as Determined by The Treating Physician
Description: The On-trial ARR was computed as the total number of relapses divided by the total number of participant years in the study period.
Time Frame: Baseline up to end of study (up to 6.5 years)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: relapses/years on study
Arm/Group | Placebo/Eculizumab | Eculizumab/Eculizumab
Number analyzed (Participants) | 41 | 78
relapses/years on study | 0.128 (0.4576) | 0.061 (0.2186)

5. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) Score
Description: Disease-related disability was measured by the EDSS. The EDSS quantifies disability in 8 Functional Systems (FS) and allows neurologists to assign a Functional System Score (FSS) in each of these. The Functional Systems are pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, cerebral, and other. The EDSS is an ordinal clinical rating scale that ranges from 0 (normal neurologic examination) to 10 (death) in half-point increments. A decrease in score indicates improvement. Baseline was defined as the last available assessment prior to the first study drug infusion in Study ECU-NMO-302.
Time Frame: Baseline, Weeks 52, 104 and 156
Population: The Extension Full Analysis Set consisted of all participants who had received at least 1 dose of eculizumab in Study ECU-NMO-302 and had a post-IP-infusion efficacy assessment. Here, Number Analyzed signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Eculizumab | Eculizumab/Eculizumab
Number analyzed (Participants) | 41 | 78
units on a scale
  Baseline | 4.34 (1.879) | 3.97 (1.736)
  Change from Baseline at Week 52: number analyzed (Participants) | 35 | 73
  Change from Baseline at Week 52 | -0.24 (0.721) | 0.01 (0.571)
  Change from Baseline at Week 104: number analyzed (Participants) | 22 | 36
  Change from Baseline at Week 104 | -0.39 (0.830) | -0.11 (0.536)
  Change from Baseline at Week 156: number analyzed (Participants) | 13 | 16
  Change from Baseline at Week 156 | -0.38 (1.003) | -0.38 (1.057)

6. Secondary Outcome: Change From Baseline in Modified Rankin Scale (mRS) Score
Description: Disease-related disability was measured by the mRS score. The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered from a neurological disability. The scale ranges from 0 (no symptoms at all) to 6 (death) in whole-point increments. A decrease in score indicates improvement. Baseline was defined as the last available assessment prior to the first study drug infusion in Study ECU-NMO-302.
Time Frame: Baseline, Weeks 52, 104 and 156
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Eculizumab | Eculizumab/Eculizumab
Number analyzed (Participants) | 41 | 78
units on a scale
  Baseline | 2.39 (1.358) | 1.88 (1.269)
  Change from Baseline at Week 52: number analyzed (Participants) | 37 | 72
  Change from Baseline at Week 52 | -0.27 (0.932) | -0.04 (0.458)
  Change from Baseline at Week 104: number analyzed (Participants) | 22 | 36
  Change from Baseline at Week 104 | -0.41 (1.182) | -0.14 (0.543)
  Change from Baseline at Week 156: number analyzed (Participants) | 13 | 16
  Change from Baseline at Week 156 | -0.62 (1.446) | -0.31 (0.602)

7. Secondary Outcome: Change From Baseline in Hauser Ambulation Index (HAI) in Participants With Abnormal Baseline Ambulatory Function
Description: The HAI evaluates gait and was used to assess the time and effort used by the participant to walk 25 feet (8 meters). The scale ranges from 0 to 9, with 0 being the best score (asymptomatic; fully active) and 9 being the worst (restricted to wheelchair; unable to transfer self independently). A decrease in score indicates improvement. Baseline is defined as the last available assessment prior to the first study drug infusion in Study ECU-NMO-302.
Time Frame: Baseline, Weeks 52, 104 and 156
Population: The Extension Full Analysis Set consisted of all participants who had received at least 1 dose of eculizumab in Study ECU-NMO-302 and had a post-IP-infusion efficacy assessment. Here, Number of Participants Analyzed signifies those participants who were evaluable for this outcome measure and Number Analyzed signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Eculizumab | Eculizumab/Eculizumab
Number analyzed (Participants) | 40 | 66
units on a scale
  Baseline | 2.83 (2.123) | 2.35 (2.257)
  Change from Baseline at Week 52: number analyzed (Participants) | 36 | 59
  Change from Baseline at Week 52 | -0.44 (1.132) | 0.08 (0.816)
  Change from Baseline at Week 104: number analyzed (Participants) | 21 | 29
  Change from Baseline at Week 104 | -0.57 (1.777) | 0.07 (1.033)
  Change from Baseline at Week 156: number analyzed (Participants) | 13 | 14
  Change from Baseline at Week 156 | -1.08 (1.706) | 0.07 (1.269)

8. Secondary Outcome: Change From Baseline in European Quality of Life (EuroQoL) 5-Dimension Visual Analog Scale (EQ-5D VAS) Health Status Score
Description: The EQ-5D is a generic, standardized participant self-administered health status instrument. EQ-5D general health status can also be measured by a visual analog scale (EQ-5D VAS). EQ-5D-VAS recorded the participant's self-rated health on a vertical visual analog scale (VAS) that allowed the participants to indicate their health state that ranged from 0 (worst imaginable) to 100 (best imaginable). Baseline is defined as the last available assessment prior to the first study drug infusion in Study ECU-NMO-302.
Time Frame: Baseline, Weeks 52, 104 and 156
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Eculizumab | Eculizumab/Eculizumab
Number analyzed (Participants) | 41 | 78
units on a scale
  Baseline | 62.00 (22.012) | 72.27 (20.941)
  Change from Baseline at Week 52: number analyzed (Participants) | 37 | 73
  Change from Baseline at Week 52 | 2.22 (13.294) | -0.78 (12.388)
  Change from Baseline at Week 104: number analyzed (Participants) | 22 | 36
  Change from Baseline at Week 104 | 0.05 (18.867) | 1.28 (11.295)
  Change from Baseline at Week 156: number analyzed (Participants) | 13 | 16
  Change from Baseline at Week 156 | 11.00 (19.374) | -4.13 (18.421)

9. Secondary Outcome: Change From Baseline in Kurtzke Visual Functional System Scores (FSS) in Participants With Abnormal Baseline Visual Function
Description: The EDSS assesses multiple Kurtzke functional systems in the context of a standard neurological exam, including visual function. The visual score ranges from 0 to 6. A score of 0 implies the participant has normal visual function. Higher scores represent worse disability. Baseline is defined as the last available assessment prior to the first study drug infusion in Study EC-NMO-302.
Time Frame: Baseline, Weeks 52, 104 and 156
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Eculizumab | Eculizumab/Eculizumab
Number analyzed (Participants) | 28 | 67
units on a scale
  Baseline | 3.75 (2.030) | 3.60 (2.031)
  Change from Baseline at Week 52: number analyzed (Participants) | 26 | 62
  Change from Baseline at Week 52 | -0.08 (0.392) | -0.06 (0.569)
  Change from Baseline at Week 104: number analyzed (Participants) | 15 | 31
  Change from Baseline at Week 104 | -0.13 (0.352) | -0.10 (0.651)
  Change from Baseline at Week 156: number analyzed (Participants) | 11 | 14
  Change from Baseline at Week 156 | 0.00 (0.000) | -0.29 (0.994)

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (up to 6.5 years)
Description: The Extension Safety Set consisted of all participants who had received at least 1 dose of eculizumab in Study ECU-NMO-302.
Groups:
- Eculizumab (Combined Total): All participants who received at least 1 dose of eculizumab in the extension study. Participants received open-label eculizumab (1200 mg) every 2 weeks starting at Week 4 and continued for up to 6.5 years.
Arm/Group | Placebo/Eculizumab | Eculizumab/Eculizumab | Eculizumab (Combined Total)
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/78 | 0/119
Serious Adverse Events (participants affected / at risk) | 14/41 | 26/78 | 40/119
Other Adverse Events (participants affected / at risk) | 40/41 | 70/78 | 110/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo/Eculizumab (N=41) | Eculizumab/Eculizumab (N=78) | Eculizumab (Combined Total) (N=119)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3) | 5 (5)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gonorrhoea (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Infective tenosynovitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Psoas abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Neuromyelitis optica spectrum disorder (Nervous system disorders) | 2 (4) | 3 (4) | 5 (8)
Optic neuritis (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Hemiparaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle spasticity (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Neuromuscular blockade (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Neuromyelitis optica pseudo relapse (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Anembryonic gestation (Pregnancy, puerperium and perinatal conditions) | 0/36 (0) | 1/74 (1) | 1/110 (1)
Catatonia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0/36 (0) | 1/74 (1) | 1/110 (1) — The N for this adverse event has been adjusted to the number of females in the study as it is a sex-specific event.
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Eculizumab (N=41) | Eculizumab/Eculizumab (N=78) | Eculizumab (Combined Total) (N=119)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 6 (7) | 9 (10)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (5) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 8 (17) | 6 (11) | 14 (28)
Constipation (Gastrointestinal disorders) | 4 (5) | 6 (7) | 10 (12)
Nausea (Gastrointestinal disorders) | 7 (17) | 3 (4) | 10 (21)
Dyspepsia (Gastrointestinal disorders) | 4 (5) | 2 (9) | 6 (14)
Toothache (Gastrointestinal disorders) | 5 (7) | 1 (1) | 6 (8)
Dental caries (Gastrointestinal disorders) | 1 (1) | 4 (5) | 5 (6)
Pyrexia (General disorders) | 6 (8) | 12 (19) | 18 (27)
Fatigue (General disorders) | 4 (13) | 7 (7) | 11 (20)
Oedema peripheral (General disorders) | 1 (1) | 4 (4) | 5 (5)
Peripheral swelling (General disorders) | 3 (4) | 2 (2) | 5 (6)
Nasopharyngitis (Infections and infestations) | 16 (35) | 13 (32) | 29 (67)
Upper respiratory tract infection (Infections and infestations) | 11 (24) | 17 (27) | 28 (51)
Urinary tract infection (Infections and infestations) | 11 (29) | 13 (30) | 24 (59)
Influenza (Infections and infestations) | 9 (14) | 10 (11) | 19 (25)
Cystitis (Infections and infestations) | 4 (6) | 5 (6) | 9 (12)
Oral herpes (Infections and infestations) | 4 (17) | 4 (4) | 8 (21)
Bronchitis (Infections and infestations) | 3 (6) | 4 (6) | 7 (12)
Herpes zoster (Infections and infestations) | 3 (3) | 2 (2) | 5 (5)
Pharyngitis (Infections and infestations) | 4 (4) | 1 (1) | 5 (5)
Periodontitis (Infections and infestations) | 0 (0) | 4 (5) | 4 (5)
Pneumonia (Infections and infestations) | 3 (4) | 1 (2) | 4 (6)
Sinusitis (Infections and infestations) | 3 (4) | 1 (4) | 4 (8)
Contusion (Injury, poisoning and procedural complications) | 6 (10) | 4 (6) | 10 (16)
Thermal burn (Injury, poisoning and procedural complications) | 3 (8) | 3 (3) | 6 (11)
Fall (Injury, poisoning and procedural complications) | 3 (14) | 0 (0) | 3 (14)
Blood pressure increased (Investigations) | 3 (3) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (13) | 15 (25) | 23 (38)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (9) | 11 (24) | 16 (33)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (13) | 7 (22) | 12 (35)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (7) | 5 (6) | 10 (13)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 5 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 5 (5)
Headache (Nervous system disorders) | 12 (34) | 15 (140) | 27 (174)
Dizziness (Nervous system disorders) | 3 (3) | 5 (7) | 8 (10)
Hypoaesthesia (Nervous system disorders) | 2 (3) | 5 (6) | 7 (9)
Paraesthesia (Nervous system disorders) | 3 (3) | 3 (4) | 6 (7)
Insomnia (Psychiatric disorders) | 3 (4) | 3 (4) | 6 (8)
Urinary incontinence (Renal and urinary disorders) | 3 (3) | 1 (1) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 5 (9) | 12 (19)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (9) | 9 (13)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5) | 6 (7)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2) | 5 (7)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (5) | 6 (8)
Dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3)
Skin lesion (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT02003144/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT02003144/SAP_001.pdf